CLINICAL TRIAL: NCT07243730
Title: Determination of the Early Postprandial Essential Amino Acid Bioavailability of Yogurt vs Milk A Randomized Controlled Clinical Trial in Healthy Volunteers - A Bioavailability Study -
Brief Title: Amino Acids in the Blood After Eating Yoghurt and Milk Proteins
Acronym: NutraFerm2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 25REX0091083
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Bioavailability of Amino Acids
Keywords: Amino acids; Yogurt; Milk

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical study in healthy participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yogurt first, Milk second (Active Comparator): All subjects will receive 2 study products on separate visits in a randomized order.
  Interventions: Other: Full fat yogurt (fermented); Other: Generic full fat pasteurized milk (non-fermented)
- Milk first, Yogurt second (Active Comparator): All subjects will receive 2 study products on separate visits in a randomized order.
  Interventions: Other: Full fat yogurt (fermented); Other: Generic full fat pasteurized milk (non-fermented)

INTERVENTIONS:
Other: Full fat yogurt (fermented) — Test
Other: Generic full fat pasteurized milk (non-fermented) — Control

SUMMARY:
Participants will visit the study site twice in a fasting state. Participants asked to consume one of the two study products in a random order. Participants will consume one serving of the study product (T = 0 minutes). Study product intake should take place within 10 minutes (+/-5 minutes). Two blood samples will be taken at baseline and then at 14 timepoints after product intake. A follow up call will take place 7 (-3/+7) days after the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 40 years at the time of (Informed Consent Form) ICF signature
2. Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
3. Signed informed consent
4. Willingness and ability to comply with the protocol
5. Judged by the Investigator to be in good health.

Exclusion Criteria:

1. Any known surgery or ongoing medical condition that interferes significantly with protein absorption and digestion, and/or gastrointestinal (GI) function in the opinion of the investigator, including but not limited to the following: phenylketonuria, pancreatitis, short bowel syndrome, inflammatory bowel disease, celiac disease, gastroesophageal reflux disease, gastric ulcer, chronic gastritis, gastrointestinal cancer, esophageal and/or gastric surgery, and any cardiovascular disease (such as hypertension, arrhythmia, or atrial fibrillation) which is not controlled with the use of medication/therapy.
2. Known renal or hepatic diseases that may interfere with protein metabolism in the opinion of the investigator, including but not limited to acute hepatitis, chronic liver disease, nephritis, cystinuria, chronic kidney disease.
3. Use of systemic medication within the past 3 weeks prior to screening which in the opinion of the investigator may influence gastric acid production and/or gastrointestinal motility or function and/or protein metabolism (e.g., antibiotics, anticonvulsants, prokinetics, antacids or gastric acid inhibitors, opioid analgesics, anticoagulants, corticosteroids, laxatives, growth hormone, testosterone, immunosuppressants, or insulin).
4. Known Diabetes Mellitus Type I or Type II, insulin resistance, or metabolic syndrome.
5. Any ongoing cancer and/or cancer treatment (except for non-melanoma skin cancer or carcinoma in situ).
6. Known anaemia.
7. A blood donation within 56 days (8 weeks) for men; or 122 days (4 months) for women; prior to the screening.
8. Any known bleeding disorder.
9. Adherence to a strict dietary regime (e.g. vegetarian/ vegan/ paleo/ ketogenic/ intermittent fasting/ high protein diet (>1.6 g/kg body weight/day)) or a weight loss program.
10. Any known allergies or intolerances to ingredients of the study product, i.e. cow's milk allergies, lactose intolerance.
11. Known pregnancy and/or lactation.
12. Current smoking / vaping / use of e-cigarette / or stopped smoking for < 1 month prior to screening (except for incidental smoking of ≤ 3 cigarettes/ e-cigarettes/ cigars/ pipes per week on average in the last month prior to screening).
13. Average alcohol use of > 21 glasses per week for men or > 14 glasses per week for women (on average during the last 6 months prior to screening).
14. Drug or medicine abuse in the opinion of the investigator.
15. Current eating disorders, e.g. anorexia nervosa, bulimia nervosa, binge eating disorder.
16. Use of protein, amino acid, or creatine supplements within 4 weeks prior to screening.
17. Known difficulties with placement of and/or blood drawings from a cannula.
18. Participation in any other clinical study with investigational or marketed products concomitantly or within four weeks before study visit 1.
19. Major medical or surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation relevant in the opinion of the investigator.
20. Investigator's uncertainty about the willingness or ability of the participant to comply with the protocol requirements.
21. Employees of Danone Global Research & Innovation Center and of the investigational site and/or their family members or relatives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incremental Area Under the Curve (iAUC ₀-₁₂₀) for Essential Amino Acids (EAA) in Blood After Ingestion of Product A or Product B | 2 hours

SECONDARY OUTCOMES:
Incremental Area Under the Curve (iAUC ₀-₃₀₀) for Essential Amino Acids in Blood After Ingestion of Product A or Product B | 5 hours
Incremental Area Under the Curve (iAUC ₀-₁₂₀) for Total Amino Acids in Blood After Ingestion of Product A or Product B | 2 hours
Incremental Area Under the Curve (iAUC ₀-₃₀₀) for Total Amino Acids in Blood After Ingestion of Product A or Product B | 5 hours
Maximum Concentration (Cmax) of Total Amino Acids and Essential Amino Acids in Blood After Ingestion of Product A or Product B | 5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- EB Medical Research, Almere Stad, Netherlands

IPD SHARING:
Plan to Share IPD: No